CLINICAL TRIAL: NCT01674257
Title: An Investigation of the Role of 18F-Sodium Fluoride and 18F-Flurodeoxyglucose PET CT and USPIO Enhanced MRI in Imaging Carotid Artery Inflammation and Mineralization.
Brief Title: Metabolic Imaging in Carotid Atherosclerosis
Acronym: MICA
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MICA-V1.3; PG/12/8/29371 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Atherosclerosis; Stroke
Keywords: Atherosclerosis; Stroke; Positron-emission tomography; Ferumoxytol; Magnetic resonance imaging; Genetics; Calcification; Inflammation; Flurodeoxyglucose F18; Radiopharmaceuticals
MeSH Terms: conditions — Atherosclerosis; Stroke; Calcinosis; Inflammation | interventions — ferumoxtran-10

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and excised carotid atheroma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Carotid Endarterectomy: Patients due to undergo carotid endarterectomy for symptomatic carotid artery stenosis will undergo an 18F-Fluoride PET/CT, an 18F-Flurodeoxyglucose PET/CT and a USPIO (ferumoxytol)-enhanced MRI scan (2 MRI scans).
  Interventions: Other: USPIO (ferumoxytol)-enhanced MRI scan; Radiation: 18f-Fluoride PET/CT scan; Radiation: 18F-Flurodeoxyglucose PET/CT scan

INTERVENTIONS:
Other: USPIO (ferumoxytol)-enhanced MRI scan — Two separate MRI scans will form this intervention. A baseline scan followed by an infusion of USPIO (ferumoxytol), followed by another MRI scan.
Radiation: 18f-Fluoride PET/CT scan
Radiation: 18F-Flurodeoxyglucose PET/CT scan

SUMMARY:
Hardening of the arteries (atherosclerosis) is a common disorder that causes heart attacks and strokes. PET CT and contrast-enhanced MRI scans are two new ways of assessing atherosclerosis. The investigators propose to perform PET CT and MRI scans on patients with hardening of the neck arteries due to undergo surgery to remove the hardened areas. The investigators will then be able to compare the hot spots found on these scans with what the investigators can see in the removed specimens under the microscope in the laboratory. This will give investigators insight into the value of PET CT and MRI as tools for assessing atherosclerosis. It will also provide the investigators with new information relating to the underlying processes that give rise to atherosclerosis and will pave the way for the future development of new treatments.

DETAILED DESCRIPTION:
Hardening of the arteries (atherosclerosis) is a very common health problem that can lead to fatal or disabling heart attacks and strokes. On many levels, it remains an incompletely understood illness.

Until relatively recently, the only way of assessing the severity of, or risk posed by, atherosclerosis was to measure the degree to which it narrowed a particular blood vessel. This method only tells part of the story; he investigators now know that frequently the 'culprit area' of atherosclerosis that causes the heart attack or stroke does not necessarily result in narrowing of the blood vessel - i.e. if the investigators only measure narrowness the investigators will miss lots of 'bad' atherosclerosis. As such, there is a pressing need to identify more sophisticated techniques of assessing the disease in order that people who are at higher risk of heart attack or stroke can be identified early and offered appropriate preventative treatment.

Techniques that provide this extra information could also significantly shorten the time it takes to get new treatments and drugs to market by providing a faster and more cost-effective way of assessing these treatments early in their development. Furthermore, in exploring new techniques that reflect more accurately what is going on within atherosclerosis in the body, deeper insight into the condition will be gained. This will in turn lead to the development of new treatments.

PET/CT scans and USPIO (a kind of tracer) enhanced MRI scans are two such techniques that demonstrate particular promise. These scanning methods not only provide more information about the composition and architecture of the atherosclerosis but can provide data about the processes (at the chemical and cellular level) that underlie the disease.

Inflammation and calcification (deposits of calcium) are two biological processes that are known to be very important in the genesis of atherosclerosis. PET/CT and USPIO enhanced MRI can detect these processes.

Most strokes and mini-strokes are caused by a narrowing in the neck artery. If a patient with mini-stroke or stroke has a narrowing (atherosclerosis) in their carotid artery they are normally offered an operation to remove the atherosclerosis (endarterectomy), the piece of atherosclerosis is then normally discarded. This scenario affords a perfect opportunity to explore new scanning techniques.

The investigators propose to explore the feasibility and value of using PET/CT (using 18F-FDG and 18F-NaF - two tracers known to highlight inflammation and calcification) and USPIO enhanced MRI to assess atherosclerosis. The investigators will do this by scanning patients who have just had a mini-stroke or minor stroke and are due to undergo endarterectomy. The investigators will then be able to define what is going on at the level of the genes and the cells that causes 'hot spots' on CT/PET and MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carotid stenosis due to undergo carotid endarterectomy.

Exclusion Criteria:

* Patients with new stroke and a modified Rankin score >3
* Chronic Kidney Disease with eGFR of <30 mL/min/1.73m2
* Pregnant women
* Poorly controlled diabetes mellitus (HbA1c > 8.5%) or diabetes mellitus requiring insulin
* Prior ipsilateral carotid intervention
* Prior neck irradiation
* Inability to tolerate the supine position
* Participation in the study would result in delay to surgery
* Psychiatric illness/social situations that would limit compliance with study requirements
* Specific contraindications to MRI (e.g. pacemaker)
* History of allergic reaction attributed to ferumoxytol or similar
* Known or suspected iron overload (genetic haemochromatosis or history of multiple transfusions)
* History of allergic reaction attributed to 18F-FDG or 18F-NaF or similar
* History of allergic reaction to iodine or iodine-based contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for carotid endarterectomy for symptomatic carotid artery stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
The Standardized Uptake Value (SUV) for 18F-Fluoride of the ipsilateral carotid artery | 1-2 days after PET/CT scan
  The mean and maximum SUV (using 18F-NaF) of the ipsilateral carotid artery will be calculated and compared to its contra lateral partner. The SUV is a validated quantitative assessment of PET radiotracer uptake.

SECONDARY OUTCOMES:
The SUV of 18F-Flurodeoxyglucose on PET/CT of the ipsilateral carotid artery | 1-2 days after PET/CT scan
  The mean and maximum SUV (using 18F-Flurodeoxyglucose) of the ipsilateral carotid artery will be calculated and compared to its contra lateral partner.
A correlation between the ipsilateral carotid SUV of 18F-Flurodeoxyglucose and tissue markers of inflammation and apoptosis. | Approximately 1 month after PET/CT scan
  Sections of excised atheroma that demonstrate uptake of 18F-Flurodeoxyglucose will be subjected to histological examination. A variety of immunohistochemical markers of inflammation and apoptosis will be quantitatively assessed for correlation with the degree of radioligand uptake. Tissue showing no radioligand uptake will be used as control.
A correlation between ipsilateral carotid SUV of 18F-Fluoride and the gene expression characteristics of excised plaque. | Approximately 1 month after the PET/CT scan
  Sections of excised atheroma that demonstrate uptake of 18F-Fluoride will be subjected to gene expression profiling. Sections of plaque that do not show uptake will be used as controls. The resulting data will be analyzed to explore the variation in gene expression between subjects and between areas of differing radioligand uptake. Genes of particular interest (either identified during expression profiling or selected beforehand) will be further studied using quantitative PCR.
A correlation between the ipsilateral carotid SUV of 18F-Fluoride and tissue markers of apoptosis and calcification. | Approximately 1 month after the PET/CT scan
  Sections of excised atheroma that demonstrate uptake of 18F-Fluoride will be subjected to histological examination. A variety of immunohistochemical markers of calcification and apoptosis will be quantitatively assessed for correlation with the degree of radioligand uptake. Tissue showing no radioligand uptake will be used as control.
The presence or absence of USPIO (ultra-small superparamagnetic particles of iron oxide) uptake on MRI (magnetic resonance image) within the ipsilateral carotid artery compared to its contralateral partner. | 1-2 days after MRI scan
  USPIOs are known to accumulate within activated macrophages in inflamed atheroma. This causes a demonstrable drop in T2* signal on MR.
A correlation between the ipsilateral carotid USPIO uptake and tissue markers of inflammation and apoptosis. | 1 month after MRI scan
  Sections of excised atheroma will be co-stained for USPIO and a variety of immunohistochemical markers of inflammation and apoptosis.
A correlation between the ipsilateral carotid USPIO uptake and gene expression characteristics of excised atheroma. | 1 month after the MRI scan
  Sections of excised atheroma that demonstrate uptake of USPIO will be subjected to gene expression profiling. Sections of plaque that do not show uptake will be used as controls. The resulting data will be analyzed to explore the variation in gene expression between subjects and between areas of differing USPIO uptake. Genes of particular interest (either identified during expression profiling or selected beforehand) will be further studied using quantitative PCR.
The ipsilateral carotid radioactivity, arterial blood radioactivity and whole blood fluoride concentration measured over time | During the 18F PET/CT scan
  The kinetics of 18F-Fluoride in atherosclerosis have not yet been defined. Using data from the PET scanner in list mode and regular arterial and venous blood sampling in 20 patients (a subset of the total) we will define a model describing the radiopharmacokinetics of 18F-Fluoride in carotid atheroma.

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, DSc, Principal Investigator — University of Edinburgh
Locations (1):
- Clinical Research Imaging Centre, Edinburgh, United Kingdom